CLINICAL TRIAL: NCT01484704
Title: The Significance of MRI in the Development of Diagnostics and Treatment of Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 63/180/2010
Record Dates: First submitted 2011-11-30; First posted 2011-12-02 (Estimated); Last update posted 2011-12-02 (Estimated); Status verified 2011-11

CONDITIONS: Mammary Ductal Carcinoma
Keywords: Carcinoma ductale mammae
MeSH Terms: conditions — Carcinoma, Ductal, Breast

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- No treatment
- MRI

SUMMARY:
The purpose of this study is to determine how MRI changes the treatment and diagnostics of ductal breast cancer. 100 women with newly diagnosed breast cancer will participate the study.

ELIGIBILITY:
Inclusion Criteria:

* Tumor size less than 2cm
* Ductal carcinoma unifocal

Exclusion Criteria:

* Previous breast cancer

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Newly diagnosted breast cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-02

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital of Turku, Turku, Finland